CLINICAL TRIAL: NCT03024086
Title: Efficacy and Safety of DWJ1252 in the Treatment of Functional Dyspepsia: A Multicenter, Randomized, Double-blind, Active-controlled Study (PART 1)
Brief Title: Efficacy and Safety of DWJ1252 in the Treatment of Functional Dyspepsia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1252002
Record Dates: First submitted 2016-12-29; First posted 2017-01-18 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DWJ1252 (Experimental): DWJ1252 + Placebo of Gasmotin
  Interventions: Drug: DWJ1252
- Gasmotin (Active Comparator): Gasmotin + Placebo of DWJ1252
  Interventions: Drug: Gasmotin

INTERVENTIONS:
Drug: DWJ1252 — DWJ1252 and Placebo of Gasmotin
  Arms: DWJ1252
Drug: Gasmotin — Gasmotin and Placebo of DWJ1252
  Arms: Gasmotin

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of DWJ1252 in treatment of Functional Dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Male of female of at least 19 years old
* Patient with functional dyspepsia met the ROME III criteria

Exclusion Criteria:

* Patients with previous gastrointestinal surgery
* Patients with history of gastrointestinal bleeding, mechanical obstruction, perforation
* Patients with history of gastrointestinal cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
The change from baseline in GIS (Gastrointestinal Symptom Score) | At 4 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No